CLINICAL TRIAL: NCT06713083
Title: Physical Activity in Bed Rest Hospitalized High-Risk Pregnant Women. A Pilot Study
Brief Title: Physical Activity in Bed Rest Hospitalized High-Risk Pregnant Women
Acronym: BedRest
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Montse Palacio (Other)
Responsible Party: Sponsor-Investigator, Montse Palacio, Head of Maternal Medicine Department, Hospital Clinic of Barcelona
Organization: Hospital Clinic of Barcelona (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Bed RestPregnancy
Record Dates: First submitted 2024-11-22; First posted 2024-12-03 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Bed Rest; Pregnancy; Pregnancy Complications
Keywords: Bed rest; Pregnancy complications; Pregnancy; Hospitalization; Exercise
MeSH Terms: conditions — Pregnancy Complications; Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: This study follows a parallel assignment model, where participants are randomized into two distinct groups. One group will follow a specifically designed exercise program tailored for individuals on bed rest during high-risk pregnancy, while the other group will receive standard care without structured physical activity. The intervention group will perform daily resistance and strength exercises adapted for execution while in bed. The control group will serve as a comparison to evaluate the impact of the exercise program on physical and emotional health, quality of life, and sleep during hospitalization. Randomization ensures unbiased allocation, and both groups will be monitored simultaneously throughout the study duration.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise group (Experimental): Pregnant women admitted in the Maternal Intermediate Care Unit who will follow the standard management for its complication and will follow a specific designed exercise program.
  Interventions: Other: Exercise
- Non-exercise group (No Intervention): Pregnant women admitted in the Maternal Intermediate Care Unit who will follow the standard management for its complication

INTERVENTIONS:
Other: Exercise — Specifically designed and structured exercise program (based on resistance/strength, designed to be executed in bed or minimal mobility). It is an adaptation from the exercise program described by Brun CR et al (Brun CR, Shoemaker JK, Bocking A, Hammond JA, Poole M, Mottola MF. Bed-rest exercise, activity restriction, and high-risk pregnancies: a feasibility study. Applied Physiology, Nutrition, and Metabolism. 2011;36(4):577-582).
  Arms: Exercise group

SUMMARY:
This pilot study aims to evaluate the impact of a specifically designed exercise program for hospitalized high-risk pregnant individuals on bed rest. The exercise program, focused on resistance and strength training, is adapted for execution while in bed and seeks to address physical and emotional health challenges during hospitalization. The study will compare outcomes between participants who follow the exercise program and those receiving standard care. Primary outcomes include physical and emotional health parameters, quality of life, and sleep quality. Secondary outcomes focus on feasibility, adherence, and participant satisfaction. This research addresses the gap in physical activity guidelines for pregnant individuals on bed rest and explores the potential benefits of exercise to improve maternal well-being and postpartum recovery.

DETAILED DESCRIPTION:
This study investigates the feasibility and potential benefits of a specifically designed exercise program for hospitalized high-risk pregnant individuals on bed rest. The program includes resistance and strength exercises tailored to be safely performed while in bed, aiming to counteract the physiological and psychological deconditioning associated with prolonged inactivity during hospitalization.

Prolonged bed rest during pregnancy, often prescribed for high-risk conditions, can result in muscle atrophy, reduced cardiovascular capacity, and psychological distress, including anxiety, stress, and depression. Despite the known adverse effects of inactivity, there is limited evidence on structured exercise programs for this population. This pilot study seeks to fill that gap by testing an intervention designed to mitigate these negative outcomes.

Participants will be randomized into two groups: an exercise group (EG) and a no-exercise group (NEG). The EG will perform daily supervised exercises, lasting approximately 30 minutes, under the guidance of trained staff. The NEG will follow standard care without structured physical activity. The study evaluates physical health parameters (e.g., activity levels, muscle strength), mental health outcomes (e.g., anxiety, depression, stress), sleep quality, and quality of life. Secondary objectives include assessing program feasibility, recruitment rates, adherence, and participant satisfaction.

Data collection will include validated self-reported questionnaires, wearable devices (accelerometers), and clinical measures. Key endpoints will be compared between groups at regular intervals during hospitalization and at six weeks postpartum.

This pilot randomized controlled trial aims to generate knowledge on the acceptability, safety, and preliminary effectiveness of bed-rest exercise programs in high-risk pregnancies, with the goal of informing future larger-scale studies and addressing an unmet need in maternal care.

ELIGIBILITY:
Inclusion Criteria:

* Maternal age of 18 or more
* Delivery not expected within 1 week after recruitment.
* Language ability to understand the study.
* Informed consent signed.

Exclusion Criteria:

* Fetal death
* Severe mental health disorders and substance abuse disorders.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-02-26 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Physiological parameters: Time spent in moderate or vigorous activity | At enrollment, weeks 1 to 6 (if not delivered), at delivery, 6 weeks post-partum
  Time spent in moderate or vigorous activity (in minutes, summarized as average per day).
Physiological parameters: Total physical activity | At enrollment, weeks 1 to 6 (if not delivered), at delivery, 6 weeks post-partum
  Total physical activity (average per day in mG).
Physiological parameters: Handgrip strength test. | At enrollment, weeks 1 to 6 (if not delivered), at delivery, 6 weeks post-partum
  Handgrip strength test (in kg, adjusted for gender and age).
Physiological parameters: Calf Circumference measurement | At enrollment, weeks 1 to 6 (if not delivered), at delivery, 6 weeks post-partum
  Calf Circumference measurement (in cm, adjusted for gender and age).
Mental health/emotional parameters: GAD-7 | At enrollment, weeks 2, 4 and 6 (if not delivered), at delivery, 6 weeks post-partum
  GAD-7: Generalized Anxiety Disorder assessment scale (score ranging from 0 to 21). The higher the results, higher is the severity of anxiety.
Mental health/emotional parameters: Perceived Stress Scale (PSS-10) | At enrollment, weeks 2, 4 and 6 (if not delivered), at delivery, 6 weeks post-partum
  Perceived Stress Scale (PSS-10) (score ranging from 0 to 40). The higher the results, higher is the perception of stress.
Mental health/emotional parameters: Edinburg Postpartum Depression Scale | At enrollment, weeks 2, 4 and 6 (if not delivered), at delivery, 6 weeks post-partum
  Edinburg Postpartum Depression Scale (EPDS) (score -ranging from 0 to 30- and percentage of score ≥9). The higher the total score, more intense is the emotional stress.
Sleep cycle and Quality of life parameters: Sleep average per night | At enrollment, weeks 2, 4 and 6 (if not delivered), at delivery
  Sleep average per night (in minutes)
Sleep cycle and Quality of life parameters: Insomnia Severity Index (ISI) | At enrollment, weeks 2, 4 and 6 (if not delivered), at delivery
  Insomnia Severity Index (ISI) (score -ranging from 0 to 28- and percentage of score ≥8). Teh higher the score, the higher the severity of insomnia.
Sleep cycle and Quality of life parameters: WHOQOL-BREF score | At enrollment, weeks 2, 4 and 6 (if not delivered), at delivery
  Abbreviated version of the World Health Organization Quality of Life Assessment scale (WHOQOL-BREF) (score ranging from 0 to 100). The higher the score, better is the perception of quality of life.
Feasibility evaluation of the implementation of the exercise program: Time needed to recruit sample size | Through study completion, an average of 6 months
  Time needed to recruit sample size (in days)
Feasibility evaluation of the implementation of the exercise program: Number of women who declined to participate in the study | Through study completion, an average of 6 months
  Number of women who declined to participate in the study
Feasibility evaluation of the implementation of the exercise program: Number of women who give up participation in the study | Through study completion, an average of 6 months
  Number of women who give up participation in the study
Feasibility evaluation of the implementation of the exercise program: Adherence to the program | Through study completion, an average of 6 months
  Adherence to the program (number of days of actual performance of the exercise program while admitted)
Satisfaction evaluation | At delivery
  A questionnaire made specifically for the case evaluating different domains (length of the sessions, hardness of the sessions, daily repetition of the sessions, difficulty in particular exercises, willingness to repeat in case of re-admission, overall satisfaction to be included in the program) - Likert scale (1 to 5, being 1 not satisfied at all, and 5 highly satisfied).

SECONDARY OUTCOMES:
Baseline Maternal and fetal characteristics: Evaluation of physical activity (GAQ-P questionnaire) | At enrollment
  Evaluation of physical activity using the Get Active Questionnaire for Pregnancy. The questionnaire self-classifies how often and for how long she is engaged in physical activity of a light, moderate or vigorous intensity. Also, it addresses the question whether the woman should speak to her Obstetric Health Care Provider before beginning or continue to be physically active.
Baseline Maternal and fetal characteristics: Maternal age | At enrollment
  Maternal age (in years)
Baseline Maternal and fetal characteristics: Maternal weight | At enrollment
  Maternal weight (in kg)
Baseline Maternal and fetal characteristics: Ethnic group | At enrollment
  Ethnic group classified as:
  * White/European
  * Hispanic/latin American
  * Black/African Americans
  * Arabic
  * Asian
Baseline Maternal and fetal characteristics: Gestational age at recruitment | At enrollment
  Gestational age at recruitment (in weeks + days)
Baseline Maternal and fetal characteristics: Twin pregnancy | At enrollment
  Twin pregnancy (yes/no)
Baseline Maternal and fetal characteristics: Fetal growth percentile at admission | At enrollment
  Fetal growth percentile at admission (customized for gender and multiplicity)
Baseline Maternal and fetal characteristics: Medical condition that justifies hospital admission | At enrollment
  Medical condition that justifies hospital admission (hypertensive disorders, preterm labor, rupture of membranes, antepartum bleeding, others)
Baseline Maternal and fetal characteristics: Musculoskeletal limitations | At enrollment
  Musculoskeletal limitations (injuries or pathologies) (yes/no and description)
Maternal and fetal characteristics during hospital admission: Medication while admitted | At enrollment, weeks 1 to 6 (if not delivered), at delivery, 6 weeks post-partum
  Medication while admitted (antihypertensive treatment, tocolysis, magnesium sulphate, antibiotics, corticosteroids, others)
Maternal and fetal characteristics during hospital admission: Length of stay in the intermediate care unit | At enrollment, weeks 1 to 6 (if not delivered), at delivery, 6 weeks post-partum
  Length of stay in the intermediate care unit (in days)
Maternal and fetal characteristics during hospital admission: Length of hospital admission | At enrollment, weeks 1 to 6 (if not delivered), at delivery, 6 weeks post-partum
  Length of hospital admission (in days)
Maternal and fetal characteristics during hospital admission: Fetal CTG | At enrollment, weeks 1 to 6 (if not delivered), at delivery, 6 weeks post-partum
  Fetal CTG description
Maternal and fetal characteristics during hospital admission: Diet during the admission | At enrollment, weeks 1 to 6 (if not delivered), at delivery, 6 weeks post-partum
  Diet during the admission (in Kcal and special needs)
Maternal and fetal characteristics during hospital admission: Daily fluid intake | At enrollment, weeks 1 to 6 (if not delivered), at delivery, 6 weeks post-partum
  Daily fluid intake (in mL)
Perinatal outcomes: Gestational age at delivery | At delivery and 6 weeks post-partum
  Gestational age at delivery (in weeks + days)
Perinatal outcomes: Birthweight | At delivery and 6 weeks post-partum
  Birthweight (in grams) and percentile
Perinatal outcomes: SGA/growth restriction | At delivery and 6 weeks post-partum
  SGA/growth restriction (yes/no) and classification, if any
Perinatal outcomes: Mode of delivery | At delivery and 6 weeks post-partum
  Mode of delivery (spontaneous, assisted, cesarean section)
Perinatal outcomes: Composite adverse maternal outcome | At delivery and 6 weeks post-partum
  Composite adverse maternal outcome (yes/no considering any of the following: re-intervention, endometritis, infection of surgical wound, curettage, admission to intensive care unit, hysterectomy, need for transfusion, postpartum hemorrhage requiring medication other than oxytocin or ergometrine, maternal sepsis, death)
Perinatal outcomes: Neonatal admission to neonatal intensive care unit | At delivery and 6 weeks post-partum
  Neonatal admission to neonatal intensive care unit (yes/no)
Perinatal outcomes: Composite adverse neonatal outcome | At delivery and 6 weeks post-partum
  Composite adverse neonatal outcome: (yes/no considering any of the following: respiratory morbidity - respiratory distress syndrome or transient tachypnea - requiring intubation, moderate-severe bronchopulmonary dysplasia, intraventricular hemorrhage grade III-IV, early-onset sepsis, periventricular leukomalacia, necrotizing enterocolitis, retinopathy requiring laser, fetal or neonatal death)
Perinatal outcomes: Breastfeeding rates | At delivery and 6 weeks post-partum
  Breastfeeding rates

CONTACTS AND LOCATIONS:
Overall Officials: Montse Palacio, MD, PhD, Principal Investigator — Head of Maternal Medicine Department
Locations (1):
- Hospital Clínic de Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No
This is a pilot study designed to evaluate the feasibility and preliminary outcomes of the intervention. As such, no data-sharing plan has been developed. The focus of this study is to generate initial findings to inform the design of future larger-scale studies, where a detailed data-sharing plan may be established.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-07-31): https://cdn.clinicaltrials.gov/large-docs/83/NCT06713083/Prot_SAP_000.pdf